CLINICAL TRIAL: NCT04651452
Title: A Value Affirmation Intervention for Physical Symptoms and Medication Adherence in Breast Cancer Patients Taking Aromatase Inhibitors
Brief Title: Writing Interventions in Breast Cancer Patients Taking Aromatase Inhibitors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Creswell, Dr. J. David Creswell, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1R01CA236860-01A1 (NIH); 1R01CA236860-01A1 (NIH)
Record Dates: First submitted 2020-11-06; First posted 2020-12-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Aromatase Inhibitors; Value Affirmation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participant and their care provider, who prescribes their aromatase inhibitor, will remain masked to which writing condition (self-affirmation or reflective journaling) the participant is randomized into. The outcomes assessor will remain masked to which condition the participants will complete. However, the experimenter will help set up the participant's online content and, therefore, will not be masked to the writing condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Value Affirmation (Active Comparator): Participants in the value affirmation condition will complete six writing prompts regarding their personal values over the course of six months. For example, participants will be given a list of values and will be asked to rate them in order of importance within their own lives and write about a time when their top value was particularly important. Participants will write for about ten minutes each session. The intervention tasks will be completed on a secure, online website that each individual participant will be emailed a link to. Participants can also receive paper copies via postal mail if they prefer.
  Interventions: Behavioral: Value Affirmation
- Reflective Journaling (Active Comparator): Participants in the reflective journaling condition will complete six writing prompts over the course of six months. However, the reflective journaling condition will be writing about values that are not important to them and discuss why they could be important to others. In other tasks, they will write about aspects of daily life (e.g. morning routine). Participants will write for about ten minutes each session. The intervention tasks will be completed on a secure, online website that each individual participant will be emailed a link to. Participants can also receive paper copies via postal mail if they prefer.
  Interventions: Behavioral: Reflective Journaling

INTERVENTIONS:
Behavioral: Value Affirmation — Participants will complete writing tasks regarding their personal values.
  Arms: Value Affirmation
Behavioral: Reflective Journaling — Participants will complete writing tasks regarding their least important values and discuss why they may be important to others. They will also describe aspects of daily life.
  Arms: Reflective Journaling

SUMMARY:
Aromatase inhibitors are a powerful medication for reducing the risk of recurrence and increasing survival in postmenopausal breast cancer patients. However, these medications can lead to intolerable side effects, poor medication adherence, and increased stress levels. This project's broad objective is to assess whether an intervention can improve medication adherence and reduce physical symptoms and stress in breast cancer patients prescribed aromatase inhibitors. Participants will be randomly assigned to a values affirmation or reflective journaling condition. Interventions will be writing-based, one essay per month for six months. Physical symptoms and perceived stress will be assessed at baseline, post-intervention (one month after the intervention), and follow-up (six months from the post-intervention assessment and seven months after the end of the intervention). Furthermore, an electronic pill bottle will continuously assess daily compliance so that medication adherence rates during the intervention, post-intervention, and follow-up can be calculated.

DETAILED DESCRIPTION:
A sample of 250 participants will be recruited and randomly assigned to either the value affirmation (N=125) or reflective journaling (N=125) condition. Participants will complete baseline measures of physical symptoms, perceived stress, and other covariates. They will also be given an electronic pill bottle that will record whether they have daily opened and closed the bottle, signifying adherence to their prescribed medication regime. This pill bottle will sync to an online dashboard. Participants in both conditions will complete a brief essay online (or via paper and pencil for those who prefer or do not have internet access) every month for six months. Value affirmation condition essays will include prompts about important, core personal values. Reflective journaling essays will have prompts that do not include any core personal value content but ask participants, in part, to write about typical daily routines. Following the conclusion of the intervention, participants will report on their levels of perceived stress and physical symptoms. Six months following the post-intervention assessment, participants will again report their perceived stress levels and physical symptoms. A sample size of 250 has been selected for feasibility and because this sample size provides at least 80% power to detect differences for all three outcomes of interest.

A sub-study will be conducted on 80 of these participants who will complete their 3rd essay prompt in an fMRI scanner. In the scan session, participants will also complete a stress reactivity task. The sub-study will allow examination of the neural mechanism of value affirmation and reflective journaling to determine whether these neural mechanisms lead to enhanced medication adherence rates and reductions in stress and physical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis
* Prescribed an aromatase inhibitor within four weeks of enrollment or anticipates being prescribed one in the future
* Intention to take the prescribed aromatase inhibitor
* Fluency in English
* Own a smartphone that can support downloaded apps

Exclusion Criteria for fMRI component only:

* Have implanted metal
* Have an implanted electronic medical device
* Have an IUD that contains metal
* Are currently pregnant
* Have a history of claustrophobia
* Weigh more than 300 pounds

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Symptoms | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Breast Cancer Prevention Trial Symptom Checklist is a 43 item self-report of physical symptoms specific to breast cancer treatment. Participants rate how bothered they were by each symptom in the last 4 weeks on a five-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Item 43 is an open response question that asks participants to indicate and rate any additional symptoms they may be experiencing. Component symptom scale scores (e.g. musculoskeletal pain, cognitive problems, weight problems) will be determined by calculating the average score of the items that make up each scale. The symptom scale scores will range from 0 to 4. A total score for all the items will be calculated by adding the scores across all symptoms. Thus, the total scores will range from 0 to 172, with higher scores reflecting greater symptom severity.
Change in Perceived Stress | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The 10-item Perceived Stress Scale is a self-reported assessment of perceptions of stress over the past month. Total scores range from 0 to 40, with higher scores indicating higher levels of perceived stress.
Change in Medication Adherence | Change in adherence assessed daily, throughout 1-year participation in the study
  Participants will receive an electronic pill bottle that syncs over the internet in real-time to indicate when a participant opens and closes the bottle. This gives a daily record of whether the participant took their medication.
Change in Self-Reported Medication Adherence | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The NIH PROMIS Medication Adherence Scale (PMAS) is a 12-item scale that will be used to assess self-reported adherence behaviors and understand why a participant may be non-compliant or discontinue their medication with items that, in part, focus on one's attitude and experience with the medication of interest. Certain items are modified to reference aromatase inhibitors.
Health-Related Quality of Life in Breast Cancer Patients as assessed by the Functional Assessment of Cancer Therapy - Breast Cancer | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Functional Assessment of Cancer Therapy - Breast Cancer is an instrument used to assess health-related quality of life in breast cancer patients through five domains comprised of 37 items. Participants respond to each item on a five-point Likert scale. The domains include physical well-being (score ranging from 0 to 28), social/family well-being (score ranging from 0 to 28), emotional well-being (score ranging from 0 to 24), functional well-being (score ranging from 0 to 28), and the breast cancer subscale (score ranging from 0 to 40). A total score for the instrument, ranging from 0 to 148, is calculated by summing the five domain subscale scores. Higher scores are reflective of a better quality of life.
Neural Activity to the Affirmation Task | One session, midway through intervention
  Participants will complete an fMRI scan while engaging with a values affirmation or a reflective journaling task. We will specifically assess neural reward response during the task assigned compared to a control comparison condition.
Neural Activity to Stressful Task | One session, midway through intervention
  Participants will complete an fMRI scan while engaging with a stressful and socially evaluative math task designed to give participants feedback that suggests they are not performing well compared to their peers. We will specifically assess neural threat response during this task and compare those who complete the value affirmation task before the math task to those who complete the reflective journaling task prior to the math task.
Functional Neural Activity to Positive Stimuli | One session, midway through intervention
  Functional neural activity to a task displaying positive vs. neutral images. Analyses will focus on a within-subject analysis for each group, as well as between-subject analyses focusing on differences in neural reward activation to positive images for self-affirmation vs. reflective journaling. ROI and connectivity analyses will focus on the reward network. Correlations with changes in included questionnaires and medication adherence will also be assessed.
Functional Neural Activity to Negative Stimuli | One session, midway through intervention
  Functional neural activity to a task displaying negative vs. neutral images. Analyses will focus on a within-subject analysis for each group, as well as between-subject analyses focusing on differences in neural activation to negative images for self-affirmation vs. reflective journaling. ROI and connectivity analyses will focus on the threat/salience network. Correlations with changes in included questionnaires and medication adherence will also be assessed.
Change in Bodily Pain as assessed by the RAND 36-Item Health Survey 1.0 | Change from baseline to 1-month post-intervention and 7 months post-intervention
  We will utilize two questions from the RAND 36-Item Health Survey 1.0 that comprise the questionnaire's bodily pain component. The bodily pain component score is calculated by taking the average of the two pain items, which each have a range of 0 to 100. The component score also ranges from 0 to 100, where a lower score is indicative of a higher pain impact.

SECONDARY OUTCOMES:
Change in Recovery from Stress | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Brief Resilience Scale is a six-item instrument that will be used to assess one's ability to recover from stress. A final score for the instrument, which ranges from 1 to 5, is determined by taking the average of the six items that comprise the instrument. Scores ranging from 1 to 2.99 indicate low resilience, 3 to 4.3 signify normal resilience, and scores 4.31 to 5 reflect high resilience.
Change in Gratitude | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Gratitude Questionnaire-Six Item Form will be used to assess one's proneness to experience gratitude in daily life. Total scores for the instrument range from 6 to 42 where a higher score reflects a more grateful disposition.
Change in Well-Being as assessed by the Mental Health Continuum Short Form for Adults | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Mental Health Continuum Short Form for adults will be used as a measure of well-being. The instrument measures each facet of well-being: emotional, psychological, and social. The emotional well-being component score ranges from 0 to 15, the psychological well-being score ranges from 0 to 30, and the social well-being score ranges from 0 to 25. A total score is determined by calculating the sum of all items. The total score ranges from 0 to 70, with a higher score signifying a higher level of well-being.
Change in Depression Severity | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Patient Health Questionnaire is a nine-item instrument that will be utilized as a brief measure of depression severity. A total score ranges from 0 to 27 and is calculated by adding each of the nine items' scores. A higher total score signifies more severe depression levels.
Change in Engagement of Enjoyable Activities as assessed by the Pittsburgh Enjoyable Activities Test | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Pittsburgh Enjoyable Activities Test is a brief, ten-item measure that will be used to assess the frequency of a participant's engagement in various activities on a scale of 0 (never) to 4 (every day). A total score ranges from 0 to 40 where a higher score reflects the increased frequency of participation in enjoyable activities.
Change in Physical and Mental Fatigue | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Pittsburgh Fatigability Scale is a self-report questionnaire that assesses one's physical and mental fatigue in relation to activities with specific intensities and durations. Mental and physical fatigue component scores range from 0 to 50 and are determined by adding the scores of the items within the components. A higher score reflects a greater perceived physical/mental fatigability.
Change in Sleep Measures | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Pittsburgh Sleep Quality Index will be used to obtain self-reported ratings of sleep. The instrument contains numerous sleep-related components, all with score ranges from 0 to 3. A higher "subjective sleep quality" component score signifies poor sleep quality. A higher "sleep latency" component score signifies increased sleep latency. An increased "sleep duration" component score signifies decreased sleep duration. A greater "sleep efficiency" component score reflects decreased efficiency. A higher "sleep disturbance" component score represents higher levels of sleep disturbance. A greater "use of sleep medication" component score signifies increased sleep medication use. A higher "daytime dysfunction" component score reflects increased daytime dysfunction. Finally, a global score is determined by calculating the sum of the seven component scores. The global score ranges from 0 to 21, where a higher score signifies decreased sleep quality.
Change in Positive and Negative Emotional Style | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Positive and Negative Emotional Style instrument is a twelve-item measure of emotional style which asks participants how accurately six positive and six negative adjectives describe how they felt during the past day. Positive and negative emotional style component scores are determined by calculating the sum of the adjective ratings within each component. Component scores range from 0 to 24, with a high score signifying increased positive and negative mood on the respective scales.
Change in Self-Esteem | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Rosenberg Self Esteem Scale is a ten-item instrument that assesses global self-esteem. A total score is determined by calculating the sum of the item scores. The range of total scores is 10 to 40. Higher total scores reflect higher self-esteem.
Changes in Perceived Social Support | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Social Provisions Scale is a twenty-four-item measure of perceived social support that asks participants to think about the support they receive in current relationships. The six-component scores (attachment, social integration, reassurance of worth, reliable alliance, guidance, opportunity for nurturance) are determined by adding the scores of the items that comprise each component's scale. Component scores range from 4 to 16. A total score can be calculated by summing all of the items in the scale. The total scale score ranges from 4 to 96, with higher scores indicating increased levels of perceived support.
Change in Perceived Stress | Change over the 6-month duration of the intervention, measured each month
  The 4-item Perceived Stress Scale is a self-reported assessment of perceptions of stress over the past month. Total scores range from 0 to 16, with higher scores indicating higher levels of perceived stress.
Change in Spontaneous Self-Affirmation | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The Spontaneous Self-Affirmation Measure is an instrument that asks participants how they think about themselves when they feel threatened or anxious to assess the tendency to utilize self-affirming cognitions. Component scores are used to determine if participants focus on personal strengths and attributes, values and principles, or important social relationships. A total score, ranging from 1 to 7, is calculated by taking the average of the three component scores. A higher total score reflects an increased tendency to utilize self-affirming cognitions when one feels threatened or anxious.
Change in Loneliness | Change from baseline to 1-month post-intervention and 7 months post-intervention
  The UCLA Loneliness scale will be used to measure subjective feelings of loneliness and social isolation. A total score that ranges from 20 to 80 is calculated by summing the score of each item. A higher total score signifies increased feelings of loneliness.
Change in Self-Reported Medication Adherence | Change over 6-month duration of the intervention, measured each month
  The Basel Assessment of Adherence to Immunosuppressive Medication Scale (BAASIS) is used to assess self-reported medication adherence. Originally used to understand adherence to immunosuppressive medications, three items from the original scale will be modified to understand adherence to aromatase inhibitors in our study involving women diagnosed with breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: J. David Creswell, Ph.D, Principal Investigator — Carnegie Mellon University; Janine Dutcher, Ph.D, Study Director — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share data associated with self-reports (e.g. demographics, stress levels) and adherence by depositing the data at the Inter-University Consortium for Political and Social Research (ICPSR), which is an NIH-funded repository. All data and documentation will be de-identified and will be consistent with applicable laws and regulations. Submitted data will confirm with relevant data and terminology standards.
  This data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary study purposes. The study team agrees that the names and Institutions of persons either given or denied access to the data, and the bases for such decisions, will be summarized in the annual progress report.
  We agree to deposit and maintain the phenotypic data and secondary analysis of data (if any) at ICPSR. The repository has data access policies and procedures consistent with NIH data sharing policies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study team agrees to deposit outcome data into the ICPSR repository three years after the end of the grant period.
Access Criteria: The study team agrees that we will identify where the data will be available and how to access the data in any publications and presentations that we author or co-author, as well as acknowledge the repository and funding source in any publications and presentations. We will be using the ICPSR, an NIH-funded repository with policies and procedures in place to provide data access to qualified researchers, fully consistent with NIH data sharing policies, applicable laws, and regulations.

REFERENCES:
- [Background] Ganz PA, Day R, Ware JE Jr, Redmond C, Fisher B. Base-line quality-of-life assessment in the National Surgical Adjuvant Breast and Bowel Project Breast Cancer Prevention Trial. J Natl Cancer Inst. 1995 Sep 20;87(18):1372-82. doi: 10.1093/jnci/87.18.1372. PMID 7658498
- [Background] Stanton AL, Bernaards CA, Ganz PA. The BCPT symptom scales: a measure of physical symptoms for women diagnosed with or at risk for breast cancer. J Natl Cancer Inst. 2005 Mar 16;97(6):448-56. doi: 10.1093/jnci/dji069. PMID 15770009
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cella D, Land SR, Chang CH, Day R, Costantino JP, Wolmark N, Ganz PA. Symptom measurement in the Breast Cancer Prevention Trial (BCPT) (P-1): psychometric properties of a new measure of symptoms for midlife women. Breast Cancer Res Treat. 2008 Jun;109(3):515-26. doi: 10.1007/s10549-007-9682-9. Epub 2007 Sep 13. PMID 17851765
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Mccullough ME, Emmons RA, Tsang JA. The grateful disposition: a conceptual and empirical topography. J Pers Soc Psychol. 2002 Jan;82(1):112-27. doi: 10.1037//0022-3514.82.1.112. PMID 11811629
- [Background] Keyes CL. The mental health continuum: from languishing to flourishing in life. J Health Soc Behav. 2002 Jun;43(2):207-22. PMID 12096700
- [Background] Keyes CL. Mental illness and/or mental health? Investigating axioms of the complete state model of health. J Consult Clin Psychol. 2005 Jun;73(3):539-48. doi: 10.1037/0022-006X.73.3.539. PMID 15982151
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Pressman SD, Matthews KA, Cohen S, Martire LM, Scheier M, Baum A, Schulz R. Association of enjoyable leisure activities with psychological and physical well-being. Psychosom Med. 2009 Sep;71(7):725-32. doi: 10.1097/PSY.0b013e3181ad7978. Epub 2009 Jul 10. PMID 19592515
- [Background] Glynn NW, Santanasto AJ, Simonsick EM, Boudreau RM, Beach SR, Schulz R, Newman AB. The Pittsburgh Fatigability scale for older adults: development and validation. J Am Geriatr Soc. 2015 Jan;63(1):130-5. doi: 10.1111/jgs.13191. Epub 2014 Dec 31. PMID 25556993
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cohen S, Alper CM, Doyle WJ, Treanor JJ, Turner RB. Positive emotional style predicts resistance to illness after experimental exposure to rhinovirus or influenza a virus. Psychosom Med. 2006 Nov-Dec;68(6):809-15. doi: 10.1097/01.psy.0000245867.92364.3c. Epub 2006 Nov 13. PMID 17101814
- [Background] Rosenberg, M. Society and the adolescent self-image. Princeton University Press, 2015.
- [Background] Cutrona CE, Russell DW. The provisions of social relationships and adaptation to stress. Advances in Personal Relationships. 1987;1:37-67.
- [Background] Harris, P. R., Griffin, D. W., Napper, L. E., Bond, R., Schüz, B., Stride, C., & Brearley, I.. Individual differences in self-affirmation: Distinguishing self-affirmation from positive self-regard. Self and Identity. 2019; 18(6): 589-630.
- [Background] Russell D, Peplau LA, Ferguson ML. Developing a measure of loneliness. J Pers Assess. 1978 Jun;42(3):290-4. doi: 10.1207/s15327752jpa4203_11. PMID 660402
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Stewart AL, Ware JE. Measuring Functioning and Well-Being: The Medical Outcomes Study Approach. Duke University Press; Durham, NC: 1992.
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Cohen, S. and Williamson, G. Perceived Stress in a Probability Sample of the United States. Spacapan, S. and Oskamp, S. (Eds.) The Social Psychology of Health. Newbury Park, CA: Sage, 1988.
- [Background] Peipert JD, Badawy SM, Baik SH, Oswald LB, Efficace F, Garcia SF, Mroczek DK, Wolf M, Kaiser K, Yanez B, Cella D. Development of the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) Medication Adherence Scale (PMAS). Patient Prefer Adherence. 2020 Jun 9;14:971-983. doi: 10.2147/PPA.S249079. eCollection 2020. PMID 32606615
- [Background] Vrijens B, De Geest S, Hughes DA, Przemyslaw K, Demonceau J, Ruppar T, Dobbels F, Fargher E, Morrison V, Lewek P, Matyjaszczyk M, Mshelia C, Clyne W, Aronson JK, Urquhart J; ABC Project Team. A new taxonomy for describing and defining adherence to medications. Br J Clin Pharmacol. 2012 May;73(5):691-705. doi: 10.1111/j.1365-2125.2012.04167.x. PMID 22486599